CLINICAL TRIAL: NCT01494610
Title: A Comparative Bioavailability Study to Compare the Pharmacokinetic (PK) and Pharmacodynamic (PD) Effects of Fluticasone Propionate and Salmeterol Delivered by Fluticasone Propionate/ Salmeterol Combination in a Capsule-based Inhaler and a Multi-dose Dry Powder Inhaler, in Moderate Asthma Patients and Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Patients.
Brief Title: Pharmacokinetic and Pharmacodynamic (PK and PD) Study of Fluticasone Propionate and Salmeterol Combination Product Delivered in a Capsule-based Inhaler and in a Multi-dose Dry Powder Inhaler in Moderate Asthma Patients and Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 114334
Record Dates: First submitted 2011-10-27; First posted 2011-12-19 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: safety; replicated cross-over design; pharmacodynamics; Fluticasone propionate/Salmeterol; capsule-based inhaler; COPD; asthma; multi dose dry powder inhaler; bioavailability; pharmacokinetics
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Restraint, Physical; Blood Specimen Collection; Urination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SERETIDE Rotacaps (Experimental): Fluticasone propionate (250 micrograms [ug])/Salmeterol (50 ug) combination delivered in a capsule-based inhaler
  Interventions: Drug: SERETIDE Rotacaps
- SERETIDE Diskus (Active Comparator): Fluticasone propionate (250 ug)/Salmeterol (50 ug) combination delivered in a multi-dose dry powder inhaler
  Interventions: Drug: SERETIDE Diskus
- Placebo Rotacaps (Placebo Comparator): Placebo delivered in a capsule-based inhaler
  Interventions: Drug: SERETIDE Diskus
- Placebo Diskus (Placebo Comparator): Placebo delivered in a multi-dose dry powder inhaler
  Interventions: Drug: SERETIDE Rotacaps

INTERVENTIONS:
Drug: SERETIDE Rotacaps — The study consists of four treatment periods of 10 +/- 1 days each in a cross-over fashion. Each patient will be administered SERETIDE delivered via a capsule-based inhaler (Rotacaps) twice for two treatment periods and a placebo delivered via a capsule-based inhaler (Rotacaps) twice for two treatment periods in a randomised, double-blind, double-dummy fashion. Dosing is twice daily in the morning and evening over the duration of each treatment period.
  Other Names: Placebo delivered via a capsule-based inhaler; Physical examination; adverse event (AE) and serious AE assessments; clinical laboratory safety tests (blood and urine); 12-lead electrocardiogram assessment; SERETIDE delivered via a capsule-based inhaler
  Arms: Placebo Diskus; SERETIDE Rotacaps
Drug: SERETIDE Diskus — The study consists of four treatment periods of 10 +/- 1 days each in a cross-over fashion. Each patient will be administered SERETIDE delivered via a multi-dose dry powder inhaler (Diskus) twice for two treatment periods and a placebo delivered via a multi-dose dry powder inhaler (Diskus) twice for two treatment periods in a randomised, double-blind, double-dummy fashion. Dosing is twice daily in the morning and evening over the duration of each treatment period.
  Other Names: Physical examination; adverse event (AE) and serious AE assessments; clinical laboratory safety tests (blood and urine); 12-lead electrocardiogram assessment; SERETIDE delivered via a multi-dose dry powder inhaler; Placebo delivered via a multi-dose dry powder inhaler
  Arms: Placebo Rotacaps; SERETIDE Diskus

SUMMARY:
This is a comparative bioavailability study to compare the pharmacokinetics and pharmacodynamic effects of Fluticasone propionate and Salmeterol delivered in a capsule-based inhaler versus a multi-dose dry powder inhaler in patients with moderate asthma and in patients with moderate to severe Chronic obstructive pulmonary disease (COPD).

Co-primary endpoints will be the area under the curve (AUCτ) measured for plasma Fluticasone propionate (pharmacokinetic) and the pharmacodynamic effects of Fluticasone propionate (weighted mean serum cortisol over 0-12h) on the last day of each 10 day study treatment period. Secondary endpoints will include the following pharmacokinetic parameters for both fluticasone propionate and salmeterol: AUClast, AUC(0-t), Cmax, Cmin, tmax, λz, and t1/2 as well as the pharmacodynamic effects of salmeterol (pulse rate, blood pressure, electrocardiogram [ECG], potassium and glucose) and Fluticasone propionate (urine cortisol levels). Safety (adverse events and laboratory abnormalities) will also be assessed as a secondary endpoint.

The study is a randomised, double blind, double dummy, four-period cross-over study. Approximately 60 asthma or COPD patients will be randomised. Patients meeting eligibility criteria will receive Fluticasone propionate/salmeterol 250/50mcg bid, from a capsule-based inhaler and from a multi-dose dry powder inhaler for a period of 10 days each in a randomised order. All patients will receive treatment from each device twice. To maintain the double blind, each patient will receive active treatment and placebo at the same time from two separate devices.

DETAILED DESCRIPTION:
BACKGROUND This study will evaluate the comparative bioavailability of SERETIDE delivered via the established multi-dose powder inhaler ie DISKUS/Accuhaler and a new fluticasone propionate/salmeterol capsule-based inhaler. Both formulations will be delivered at the 250/50mcg (micrograms) twice daily (bid) dose strength.

STUDY RATIONALE The fluticasone propionate/salmeterol capsule-based inhaler has been developed for administration in both asthma and Chronic obstructive pulmonary disease (COPD) patients. Therefore, both disease populations are included in this study. The study will assess the performance of the two devices with respect to systemic exposure and pharmacodynamic effects. A replicated cross-over design (four period) was chosen. This design reduces subject numbers by about 50% compared to a standard 2-period cross-over design.

OBJECTIVES Primary Objective

-To compare the performance of fluticasone propionate/salmeterol administered in a capsule-based inhaler with the multi-dose dry powder inhaler by evaluating fluticasone propionate pharmacokinetic and pharmacodynamic endpoints.

Secondary Objectives

* To compare the pharmacokinetic and pharmacodynamic effects of the salmeterol component of fluticasone propionate/salmeterol after administration from a capsule-based inhaler and from the multi-dose dry powder inhaler
* To compare the safety and tolerability of fluticasone propionate/salmeterol after administration in a capsule-based inhaler with the multi-dose dry powder inhaler.

ENDPOINTS Primary Endpoints

* Pharmacokinetic endpoint: AUCτ for fluticasone propionate (area under the plasma fluticasone propionate concentration-time curve over dosing interval) on the last day of each study treatment period (Day 10).
* Pharmacodynamic endpoint: Weighted mean serum cortisol over 12h on the last day of each treatment period (Day 10).

Secondary Endpoints

* Pharmacokinetic parameters (AUClast, AUC(0-t), Cmax, Cmin, tmax, λz, and t1/2 for fluticasone propionate and salmeterol) on the last day of each treatment period (Day 10).
* Pharmacodynamic parameters:
* Fluticasone propionate: Urine cortisol excretion (0-24h) and serum cortisol Cmin on the last day (Day 10) of each treatment period,
* Salmeterol: pharmacodynamic parameters for pulse rate, blood pressure, electrocardiogram (ECG), plasma potassium and glucose (weighted mean 0-12h and Cmax/Cmin) on the last day (Day 10) of each treatment period
* Safety and tolerability: Incidence of adverse events and laboratory abnormalities

STUDY DESIGN This is a randomised, four-period cross-over, double-blind, double-dummy study. Patients meeting eligibility criteria will receive fluticasone propionate/salmeterol 250/50 mcg bid from a capsule-based inhaler and from a multi-dose dry powder inhaler for 10 days per each treatment period in a randomised order. To maintain the double blind, each patient will receive both active treatment and placebo at the same time from two separate devices. Patients already on inhaled corticosteroid (ICS) monotherapy or combination treatment prior to randomization will stop their existing treatment and switch to treatment provided by the study-provided devices.

The study has been designed to compare the administration of fluticasone propionate/salmeterol from two inhalation devices, a capsule-based inhaler and a multi-dose dry powder inhaler. Fluticasone propionate/salmeterol administered via the multi-dose dry powder inhaler will be the reference product. Fluticasone propionate/salmeterol is being developed by GlaxoSmithKline (GSK) as a capsule-based inhaler for administration for the treatment of both asthma and COPD.

TREATMENT ASSIGNMENT Subjects will be assigned to one of two treatment sequences in accordance with the randomisation schedule Sequence ABBA (Periods 1 to 4): A: Fluticasone propionate/salmeterol from a multi-dose dry powder inhaler; B: Fluticasone propionate/salmeterol from a capsule-based inhaler; B: Fluticasone propionate/salmeterol from a capsule-based inhaler; A: Fluticasone propionate/salmeterol from a multi-dose dry powder inhaler Sequence BAAB (Periods 1 to 4): B: Fluticasone propionate/salmeterol from a capsule-based inhaler; A: Fluticasone propionate/salmeterol from a multi-dose dry powder inhaler; A: Fluticasone propionate/salmeterol from a multi-dose dry powder inhaler; B: Fluticasone propionate/salmeterol from a capsule-based inhaler.

ELIGIBILITY:
INCLUSION CRITERIA:

ALL PATIENTS:

* Available for the duration of the study and able to attend the clinic for all study visits.
* Gender: male or female

A female subject is eligible to participate if she is of:

* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the protocol allowed contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential and agrees to use one of the protocol allowed contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until they have attended the site for the follow-up visit.
* Capable of giving informed consent, which includes compliance with the study requirements and restrictions listed in the consent form.
* Body mass index between 18 and 35 kg/m2 inclusive at Screening
* Able to use the inhaler devices adequately after training
* AST and ALT < 2xULN (upper limit of normal); alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QT interval corrected for heart rate (QTc)* <450 millisecond (msec)** QTc <480 msec for patients with bundle branch block

  * either QTcB (QTc Bazzett's formula) or QTcF (QTc Fridericia's formula), machine or manual overread, males or females. The specific formula that will be used in a study should be predetermined prior to the initiation of the study. The QT correction formula used to determine inclusion and discontinuation should be the same throughout the study.

    * based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period

COPD PATIENTS:

* Diagnosis: COPD patients, defined as either Stage III to Stage IV COPD diagnosis according to GOLD criteria (Global Strategy for the Diagnosis, Management, and Prevention of COPD, updated 2009) [GOLD, 2009]. Individuals must be otherwise healthy individuals who are free from significant cardiac, gastrointestinal, hepatic, renal, haematological malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations.
* Age: 40-80 years inclusive at the time of signing the informed consent.
* Post-bronchodilator forced expiratory volume in one second (FEV1) < 50% of predicted normal values at Screening. Patients must abstain from short acting beta agonist (SABA) use for 6 hours prior to the screening visit.
* Post-bronchodilator FEV1/FVC ratio ≤ 0.70 at Screening
* An increase of less than 15% from baseline FEV1 or an absolute change of < 200ml, 30 minutes after inhalation of 400mcg of salbutamol by metered-dose inhaler (MDI) and spacer or 2.5mg by nebuliser at Screening.
* Ex smokers for at least the past 3 months with a pack history ≥10 pack years [number of pack years = (number of cigarettes per day / 20) x number of years smoked].
* COPD therapy:
* Patients on fluticasone propionate/salmeterol combination 250/50mcg bid via a multi-dose dry powder inhaler prior to the study will be allowed to remain on their treatment regimen until randomization provided all other eligibility criteria are met.
* Patients on fluticasone propionate/salmeterol combination 250/50mcg bid via a metered dose inhaler or the equivalent dose of budesonide/formoterol, 800/24mcg (total daily dose) via a turbuhaler will be switched to fluticasone propionate/salmeterol combination 250/50mcg bid via the GSK provided multi-dose dry powder inhaler for between 14 and 28 days prior to randomization.
* Patients on tiotropium in addition to ICS/LABA (long-acting beta agonist) treatment (up to a total daily dose of 500mcg fluticasone propionate or other ICS equivalent eg. 800mcg budesonide) may continue their tiotropium treatment throughout the study.
* Patients on tiotropium monotherapy will need to start treatment with fluticasone propionate/salmeterol combination 250/50mcg bid via the GSK provided multi-dose dry powder inhaler for between 14 and 28 days prior to randomization. They may continue their tiotropium treatment throughout the study.
* Patients on LABA therapy (eg. salmeterol 50mcg) will need to start treatment with fluticasone propionate/salmeterol combination 250/50mcg bid via the GSK provided multi-dose dry powder inhaler for between 14 and 28 days prior to randomization.

ASTHMA PATIENTS:

* Diagnosis: Patients with moderate asthma as defined by the Global Initiative for Asthma (GINA) guidelines at Screening. A best FEV1 of 60-85% of the predicted normal value at the Screening visit. NHANES (National Health and Nutrition Examination Survey) III predicted values will be used [Hankinson, 2009]. If a subject is recorded as having Hispanic or Latino ethnicity, then the Mexican-American equations will be used (irrespective of race). If a subject is recorded as being of African American/African Heritage race, then the African American equations will be used. If a subject is recorded as being of Asian or of Pacific Islander race, then the Caucasian formula will be used with a conversion factor of 0.88. Otherwise, the Caucasian equations will be used.
* Age: 18 and above at the time of signing the informed consent.
* Best clinic screening pre-bronchodilator FEV1 between 60 and 85% of predicted normal values (NHANES III values). Patients must abstain from SABA use for 6 hours prior to the Screening visit.
* Asthma therapy:
* Patients on fluticasone propionate/salmeterol combination 250/50mcg treatment via a multi-dose dry powder inhaler prior to the study will be allowed to remain on their treatment regimen until randomization provided all other eligibility criteria are met.
* Patients on treatment with ICS alone (up to a total daily dose of 500mcg fluticasone propionate or other ICS equivalent eg. 800mcg budesonide) will be required to switch treatment to fluticasone propionate/salmeterol combination 250/50mcg bid via the GSK provided multi-dose powder inhaler for between 14 and 28 days prior to randomization if deemed appropriate.
* Patients on treatment with budesonide/eformoterol combination (up to a total daily dose of 800/24mcg via a Turbuhaler) will be required to switch to fluticasone propionate/salmeterol combination 250/50mcg bid via the GSK-provided multi-dose powder inhaler for between 14 and 28 days prior to randomization.
* Patients on treatment with fluticasone propionate/salmeterol combination at a dose up to 250/50mcg bid via a metered dose inhaler or multi-dose dry powder inhaler (eg. 100/50mcg) will be required to switch to fluticasone propionate/salmeterol combination 250/50mcg bid via the GSK-provided multi-dose powder inhaler for between 14 and 28 days prior to randomization.

EXCLUSION CRITERIA:

ALL PATIENTS:

* Any clinically relevant medical condition or abnormality identified during the screening medical assessment and procedures, physical examination, or laboratory assessments (including clinical chemistry and haematology), which in the opinion of the GSK Medical Monitor is likely to affect the safety of the subject and/or interfere with the study procedures and outcomes.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody or positive HIV test result within 3 months of screening.
* Patients on treatment with fluticasone propionate either as monotherapy or in combination at a total daily dose higher than 500mcg or budesonide monotherapy or in combination at a total daily dose higher than 800mcg are excluded from the study
* Use of oral/injectable/depot corticosteroid for any indication within 3 months prior to the Screening visit.
* Use of intra-nasal steroids (INS). To be eligible for the study, patients on INS therapy will be required to switch to non-INS therapy at randomization.
* Patients with abnormal levels of serum cortisol at Screening
* Abuse of alcohol consumption within 12 months of the Screening visit defined by the following Australian guidelines:

Males: An average weekly intake greater than 21 units or an average daily intake greater than 3 units. Females: An average weekly intake greater than 14 units or an average daily intake greater than 2 units.

One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.

* A known or suspected history of drug abuse within 12 months of the Screening visit.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56-day period.
* Known hypersensitivity to salbutamol or any ingredient in the study medication preparation and/or history of any other drug or other allergy that, in the opinion of the GSK medical monitor and the investigator contraindicates participation of the subject
* Grapefruit or grapefruit juice containing products are excluded from 2 weeks prior to randomisation until collection of the final blood sample at treatment period 4.
* Drugs that inhibit the cytochrome P450 isoform, 3A4 (CYP3A4), are excluded from 2 weeks prior to randomisation until collection of the final blood sample at treatment period 4. CYP3A4 inhibitors include cimetidine, clarithromycin, erythromycin, ciprofloxacin, ritonavir, ketoconazole, and azole antifungals, a complete list is provided in the protocol.
* Use of prescription or non-prescription drugs, vitamins, herbal and dietary supplements, within seven days or 5 half-lives (whichever is longer) prior to the first dose of study medication, which in the opinion of the Principal Investigator, may interfere with study outcome. Specifically, calcium and vitamin D supplements and bisphosphonates are not allowed throughout the study.
* Pregnant females as determined by positive serum or urine βhCG (β-human chorionic gonadotropin) test at Screening or prior to dosing.
* Patients, who, in the opinion of the Investigator, are not able to comply with the protocol requirements.

COPD PATIENTS:

* Subjects with a respiratory disorder in addition to COPD (e.g. bronchiectasis, fibrosis) or significant co-morbidity that might affect lung function (e.g. poorly controlled heart failure, atrial fibrillation or ischaemic heart disease).
* Regular oxygen or nebulised bronchodilator therapy
* The subject has history of a respiratory infection (including sinusitis) within 4 weeks prior to the Screening visit
* Any previous lung resection surgery (eg., lung volume reduction surgery or lobectomy)

ASTHMA PATIENTS:

* Acute exacerbation of asthma requiring hospitalisation in the 6 weeks prior to the Screening visit.
* Subjects may not have used inhaled tobacco products within the past 3 months (ie. cigarettes, cigars or pipe tobacco) or have historical use of 10 pack years or more; [number of pack years = (number of cigarettes per day / 20) x number of years smoked].

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10-25 (Actual); Primary Completion 2011-06-08 (Actual); Study Completion 2011-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (2):
- GSK Investigational Site, Randwick, New South Wales, Australia
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Daley-Yates PT, Mehta R, Chan RH, Despa SX, Louey MD. Pharmacokinetics and pharmacodynamics of fluticasone propionate and salmeterol delivered as a combination dry powder from a capsule-based inhaler and a multidose inhaler in asthma and COPD patients. J Aerosol Med Pulm Drug Deliv. 2014 Aug;27(4):279-89. doi: 10.1089/jamp.2013.1040. Epub 2013 Sep 28. PMID 24074143
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- FP/Salmeterol 250/50 mcg: Sequence ABBA: Participants received fluticasone propionate (FP)/salmeterol 250/50 micrograms (mcg) twice daily via a capsule-based inhaler for two 10-day periods and via a multi-dose dry powder (MDPI) inhaler for two 10-day periods in a replicate crossover design. Participants were dosed approximately every 12 hours. Treatment was given in the sequence of ABBA in Periods 1, 2, 3, and 4 (with no washouts between periods), respectively. A, FP/salmeterol from an MDPI; B, FP/salmeterol from a capsule-based inhaler.
- FP/Salmeterol 250/50 mcg: Sequence BAAB: Participants received fluticasone propionate (FP)/salmeterol 250/50 micrograms (mcg) twice daily via a capsule-based inhaler for two 10-day periods and via a multi-dose dry powder (MDPI) inhaler for two 10-day periods in a replicate crossover design. Participants were dosed approximately every 12 hours. Treatment was given in the sequence of BAAB in Periods 1, 2, 3, and 4 (with no washouts between periods), respectively. A, FP/salmeterol from an MDPI; B, FP/salmeterol from a capsule-based inhaler.
Period: Period 1
Arm/Group | FP/Salmeterol 250/50 mcg: Sequence ABBA | FP/Salmeterol 250/50 mcg: Sequence BAAB
Started | 31 | 29
Completed | 30 | 28
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 2
Arm/Group | FP/Salmeterol 250/50 mcg: Sequence ABBA | FP/Salmeterol 250/50 mcg: Sequence BAAB
Started | 30 | 28
Completed | 30 | 28
Not Completed | 0 | 0
Period: Period 3
Arm/Group | FP/Salmeterol 250/50 mcg: Sequence ABBA | FP/Salmeterol 250/50 mcg: Sequence BAAB
Started | 30 | 28
Completed | 28 | 28
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 4
Arm/Group | FP/Salmeterol 250/50 mcg: Sequence ABBA | FP/Salmeterol 250/50 mcg: Sequence BAAB
Started | 28 | 28
Completed | 27 | 28
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- FP/Salmeterol 250/50 mcg: Participants received fluticasone propionate (FP)/salmeterol 250/50 micrograms (mcg) twice daily via a capsule-based inhaler for two 10-day periods and via a multi-dose dry powder (MDPI) inhaler for two 10-day periods in a replicate crossover design. Participants were dosed approximately every 12 hours. Treatment was given in one of two sequences in Periods 1, 2, 3, and 4 (with no washouts between periods), respectively: ABBA, BAAB. A, FP/salmeterol from an MDPI; B, FP/salmeterol from a capsule-based inhaler.
Arm/Group | FP/Salmeterol 250/50 mcg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 51.1 (18.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 44
Race/Ethnicity, Customized [Number; unit: participants]
  White-White/Caucasian/European Heritage | 56
  American Indian or Alaskan Native | 2
  African American/African Heritage | 1
  Asian-Central/South Asian Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Concentration Time Curve Over the Dosing Period (AUC[0-tau]) for FP
Description: Blood samples of participants (par.) with asthma and chronic obstructive pulmonary disease (COPD) were collected and analyzed for AUC(0-tau), a measure of the amount of drug available at target tissue (in plasma) for a fixed dosing interval (12 hours). Asthma is a disorder that causes the airways of the lungs to swell and narrow, leading to difficulty in breathing. COPD is a chronic lung disease with structural changes in lungs, leading to difficulty in breathing.
Time Frame: At pre-morning dose; 5, 10, 30 minutes post-dose (PD); and 1, 2, 4, 8, 10, and 12 hours PD on Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: Pharmacokinetic/pharmacodynamic (PK/PD) Population: all participants who received at least one dose of study medication, except for one who was identified as a full protocol violator. Participants with at least one non-missing value in the replicate observations were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Picogram hours per milliliter (pg*h/mL)
Groups:
- FP/Salmeterol From MDPI: Fluticasone propionate (FP)/salmeterol combination was administered as a powder in blister in the dose of 250/50 micrograms (mcg) twice daily (BID) via a multi-dose dry powder inhaler (MDPI) for two 10-day periods
- FP/Salmeterol From Capsule-based Inhaler: Fluticasone propionate/salmeterol combination was administered as a powder in capsule in the dose of 250/50 mcg BID via a capsule-based inhaler for two 10-day periods.
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
Picogram hours per milliliter (pg*h/mL)
  Asthma + COPD; n=57, 57 | 376.9 [337.0 to 421.6] | 573.1 [519.3 to 632.5]
  Asthma; n=33, 33 | 350.5 [296.5 to 414.4] | 559.1 [490.1 to 637.7]
  COPD; n=24, 24 | 416.4 [363.1 to 477.6] | 593.0 [505.7 to 695.4]
Statistical Analysis 1: Comparison: FP/Salmeterol From MDPI vs FP/Salmeterol From Capsule-based Inhaler; Test type: Non-Inferiority or Equivalence — Estimates of within-par. coefficient of variation for AUC(0-tau) of FP and weighted mean (0-12 h) serum cortisol from previous studies showed that a sample size of 52 par. would have approximately 90% power to demonstrate biocomparability with respect to the two co-primary endpoints. The study was powered on the analysis of asthma and COPD par. as a combined group. A two one-sided t-test procedure with α=0.05 for each one-sided test was used. Biocomparability limits of 0.8 and 1.25 were used; Ratio of adjusted geometric means = 1.508, 90% CI 2-sided [1.366 to 1.665] — Data reflect Asthma + COPD participants. The ratio of adjusted geometric means is a comparision of treatment administered by the capsule-based inhaler and the MDPI
Statistical Analysis 2: Comparison: FP/Salmeterol From MDPI vs FP/Salmeterol From Capsule-based Inhaler; Test type: Non-Inferiority or Equivalence — Estimates of within-par. coefficient of variation for AUC(0-tau) of FP and weighted mean (0-12 h) serum cortisol from previous studies showed that a sample size of 52 par. would have approximately 90% power to demonstrate biocomparability with respect to the two co-primary endpoints. The study was powered on the analysis of asthma and COPD par. as a combined group. Biocomparability limits of 0.8 and 1.25 were used; Ratio of adjusted geometric means = 1.598, 90% CI 2-sided [1.369 to 1.864] — Data reflect participants with asthma only. The ratio of adjusted geometric means is a comparision of treatment administered by the capsule-based inhaler and the MDPI
Statistical Analysis 3: Comparison: FP/Salmeterol From MDPI vs FP/Salmeterol From Capsule-based Inhaler; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 1.421, 90% CI 2-sided [1.274 to 1.584] — Data reflect participants with COPD only. The ratio of adjusted geometric means is the comparision of treatment administered by the capsule-based inhaler and the MDPI

2. Primary Outcome: Weighted Mean Serum Cortisol (SC) Over 0 to 12 Hours Post Dose
Description: Participants' blood samples were collected and analyzed for SC levels. Weighted mean SC levels are evaluted as a measure of the degree of cortisol suppression, allowing for the determination of whether differences in systemic exposure to the inhaled steroid component of two devices can be significant enough to result in the differences in the body's ability to release cortisol. Weighted means were derived by calculating the AUC over the 0-12 hour period, using the linear trapezoidal rule (statistical technique used for numerical analysis) and then dividing it by the actual time interval.
Time Frame: At pre-morning dose; 30 minutes post-dose (PD); and 1, 2, 4, 8, 10, and 12 hours PD on Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanomoles per liter (nmol/L)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
Nanomoles per liter (nmol/L)
  Asthma + COPD;n=57, 57 | 193.5 [178.7 to 209.6] | 178.3 [164.2 to 193.5]
  Asthma; n=33, 33 | 187.3 [169.1 to 207.6] | 166.6 [150.4 to 184.7]
  COPD; n=24, 24 | 202.4 [177.0 to 231.4] | 195.6 [171.1 to 223.7]
Statistical Analysis 1: Comparison: FP/Salmeterol From MDPI vs FP/Salmeterol From Capsule-based Inhaler; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 0.928, 90% CI 2-sided [0.886 to 0.971] — Data reflect Asthma + COPD participants. The ratio of adjusted geometric means is the comparision of treatment administered by the capsule-based inhaler and the MDPI
Statistical Analysis 2: Comparison: FP/Salmeterol From MDPI vs FP/Salmeterol From Capsule-based Inhaler; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 0.892, 90% CI 2-sided [0.848 to 0.939] — Data reflect participants with asthma only. The ratio of adjusted geometric means is the comparision of treatment administered by the capsule-based inhaler and the MDPI
Statistical Analysis 3: Comparison: FP/Salmeterol From MDPI vs FP/Salmeterol From Capsule-based Inhaler; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjusted geometric means = 0.966, 90% CI 2-sided [0.889 to 1.049] — [estimate comment as in outcome 1, analysis 3]

3. Secondary Outcome: Mean Plasma AUC(0-tau) and Plasma AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC[0-tlast]) for Salmeterol
Description: Blood samples of participants with asthma and COPD were collected and analyzed for AUC(0-tau) and AUC(0-tlast). AUC(0-tau) is a measure of the amount of drug available at target tissue (in plasma) for a fixed dosing interval (12 hours). AUC(0-tlast) is a measure of the plasma drug concentration from pre-dose to the last measurable concentration.
Time Frame: as for outcome 1
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg*h/mL
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
pg*h/mL
  AUC(0-tau), asthma + COPD; n=57, 57 | 300.2 [273.0 to 330.1] | 345.1 [310.8 to 383.1]
  AUC(0-tau), asthma; n=33, 33 | 305.8 [274.6 to 340.6] | 356.4 [315.4 to 402.7]
  AUC(0-tau), COPD; n=24, 24 | 292.7 [244.4 to 350.5] | 330.1 [272.1 to 400.4]
  AUC(0-t), asthma + COPD; n=57, 57 | 303.5 [277.7 to 331.7] | 345.0 [310.7 to 383.0]
  AUC(0-t), asthma; n=33, 33 | 305.2 [273.9 to 340.2] | 356.4 [315.3 to 402.7]
  AUC(0-t), COPD; n=24, 24 | 301.2 [256.9 to 353.2] | 330.0 [272.0 to 400.3]

4. Secondary Outcome: Mean AUC(0-tlast) for FP
Description: Blood samples of participants with asthma and COPD were collected and analyzed for AUC(0-tlast). AUC(0-tlast) is a measure of the plasma drug concentration from pre-dose to the last measurable concentration.
Time Frame: as for outcome 1
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg*h/mL
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
pg*h/mL
  Asthma + COPD; n=57, 57 | 380.1 [342.7 to 421.6] | 580.9 [530.2 to 636.3]
  Asthma; n=33, 33 | 355.7 [306.0 to 413.4] | 558.4 [489.6 to 636.9]
  COPD; n=24, 24 | 416.5 [363.2 to 477.6] | 613.2 [539.9 to 696.5]

5. Secondary Outcome: Mean Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) of FP
Description: Blood samples of participants with asthma and COPD were collected and analyzed for Cmax and Cmin of FP in the blood. Cmax and Cmin are used to estimate the time at which the activity of the drug will be at its maximum and minimum, respectively.
Time Frame: as for outcome 1
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: Picograms per milliliter (pg/mL)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
Picograms per milliliter (pg/mL)
  Cmax, Asthma + COPD; n= 57, 57 | 54.64 [49.70 to 60.08] | 105.79 [95.70 to 116.95]
  Cmax, Asthma; n=33, 33 | 53.66 [47.36 to 60.80] | 109.98 [95.79 to 126.27]
  Cmax, COPD; n=24, 24 | 56.02 [47.91 to 65.50] | 100.29 [86.06 to 116.87]
  Cmin, Asthma + COPD; n=57, 57 | 15.904 [14.025 to 18.035] | 21.547 [19.198 to 24.183]
  Cmin, Asthma; n=33, 33 | 13.635 [11.448 to 16.239] | 18.866 [15.979 to 22.273]
  Cmin, COPD; n=24, 24 | 19.654 [16.898 to 22.859] | 25.866 [22.703 to 29.470]

6. Secondary Outcome: Mean Terminal Phase Half-life (t1/2) for FP
Description: Blood samples of participants were collected for evaluating t1/2. The t1/2 is the time required for the plasma/blood concentration of the drug to decrease by 50% after the false equilibrium of distribution has been reached.
Time Frame: as for outcome 1
Population: PK/PD Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 54 | 55
hours
  Asthma + COPD; n=54, 55 | 6.660 [6.164 to 7.197] | 5.844 [5.416 to 6.307]
  Asthma; n=30, 32 | 5.906 [5.402 to 6.458] | 5.238 [4.789 to 5.729]
  COPD; n=24, 23 | 7.740 [6.915 to 8.663] | 6.806 [6.089 to 7.607]

7. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for FP
Description: Blood samples of participants were collected for evaluating Tmax. Tmax is a measure of the time required to reach the maximum concentration of the drug.
Time Frame: as for outcome 1
Population: PK/PD Population
Measure: Median (Full Range); unit: hours
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
hours
  Asthma + COPD; n=57, 57 | 1.045 [0.08 to 5.00] | 0.530 [0.08 to 2.04]
  Asthma; n=33, 33 | 1.000 [0.08 to 4.04] | 0.335 [0.08 to 2.04]
  COPD; n=24, 24 | 1.173 [0.17 to 5.00] | 0.673 [0.13 to 1.54]

8. Secondary Outcome: Mean Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) for Salmeterol
Description: Blood samples of participants with asthma and COPD were collected and analyzed for Cmax and Cmin of Salmeterol in the blood. Cmax and Cmin are used to estimate the time at which the activity of the drug will be at its maximum and minimum.
Time Frame: as for outcome 1
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
pg/mL
  Cmax, Asthma + COPD; n=57, 57 | 59.28 [53.45 to 65.74] | 92.27 [80.52 to 105.75]
  Cmax, Asthma; n=33, 33 | 64.97 [56.53 to 74.66] | 110.21 [94.76 to 128.19]
  Cmax, COPD; n=24, 24 | 52.26 [44.94 to 60.77] | 72.27 [57.75 to 90.45]
  Cmin, Asthma + COPD; n=57, 57 | 12.752 [11.504 to 14.134] | 14.354 [12.859 to 16.024]
  Cmin, Asthma; n=33, 33 | 12.676 [11.097 to 14.479] | 14.634 [12.806 to 16.723]
  Cmin, COPD; n=24, 24 | 12.857 [10.798 to 15.307] | 13.978 [11.464 to 17.044]

9. Secondary Outcome: Mean Terminal Phase Half-life (t1/2) for Salmeterol
Description: Blood samples of participants were collected for evaluating t1/2. t1/2 is the time required for the plasma/blood concentration of the drug to decrease by 50% after the false equilibrium of distribution has been reached.
Time Frame: as for outcome 1
Population: PK/PD Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 56 | 56
hours
  Asthma + COPD; n=56, 56 | 6.576 [6.080 to 7.112] | 7.260 [6.792 to 7.761]
  Asthma; n=32, 32 | 6.429 [6.021 to 6.865] | 7.538 [6.840 to 8.308]
  COPD; n=24, 24 | 6.776 [5.727 to 8.018] | 6.905 [6.309 to 7.558]

10. Secondary Outcome: Tmax for Salmeterol
Description: as for outcome 7
Time Frame: as for outcome 1
Population: PK/PD Population
Measure: Median (Full Range); unit: hours
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
hours
  Asthma + COPD; n=57, 57 | 0.750 [0.08 to 6.50] | 0.080 [0.08 to 6.50]
  Asthma; n=33, 33 | 0.335 [0.08 to 6.50] | 0.080 [0.08 to 1.04]
  COPD; n=24, 24 | 1.000 [0.08 to 2.00] | 0.080 [0.08 to 6.50]

11. Secondary Outcome: Mean Urine Cortisol Excretion Over 0 to 24 Hours Post Dose for FP
Description: Urine samples of participants were collected to evaluate urine cortisol excretion over 0-24 hours post treatment dose. A 24-hour urine cortisol sample was used to measure the total amount of cortisol excreted in urine in 24 hours. Any differences in systemic exposure as a result of the absorbed steroid component of the two differing inhaled devices should also result in differences in the amount of cortisol excreted in the urine.
Time Frame: 0-24 hours post dose on Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: nmol
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
nmol
  Asthma + COPD; n=57, 57 | 63.53 [56.71 to 71.17] | 59.66 [51.45 to 69.18]
  Asthma; n=33, 33 | 72.86 [62.97 to 84.32] | 66.28 [55.25 to 79.51]
  COPD; n=24, 24 | 52.62 [44.77 to 61.83] | 51.62 [40.16 to 66.35]

12. Secondary Outcome: Serum Cortisol Minimum (Cmin) for FP
Description: Blood samples of participants were collected for the evaluation of minimum serum cortisol. Any differences in systemic exposure as a result of the absorbed steroid component of the two differing inhaled devices should also result in differences in serum cortisol concentrations.
Time Frame: Day 10 of each study period (Periods 1-4); Study Day 10 (+/-1) (reference day is Study Day 1 or Randomization day), Period 1; Study Day 20 (+/-1), Period 2; Study Day 30 (+/-1), Period 3; Study Day 40 (+/-1), Period 4
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
nmol/L
  Asthma + COPD; n=57, 57 | 88.6 [77.9 to 100.8] | 79.6 [69.0 to 91.7]
  Asthma; n=33, 33 | 79.8 [67.0 to 95.0] | 70.0 [57.8 to 84.7]
  COPD; n=24, 24 | 102.4 [85.0 to 123.3] | 94.9 [77.1 to 116.8]

13. Secondary Outcome: Weighted Mean Over 0 to 4 Hours Post Dose of Heart Rate for Salmeterol
Description: The heart rate (number of heartbeats per unit of time, typically expressed as beats per minute [bpm]) of the participants was monitored for evaluating the weighted mean over the course of 0 to 4 hours post dose. The Capsule-MDPI difference for heart rate was calculated for each participant, and the weighted mean value from the time of the morning dose on Day 10 to 4 hours post dose was calculated. The weighted mean was calculated by using all values at the indicated timepoint contributing to the calculation of the mean but with different weightage.
Time Frame: At pre-morning dose; 15, 30, 60, 90 minutes post-dose (PD); and 2, 4, 8, 10, and 12 hours PD on Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: PK/PD Population
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
bpm
  Asthma + COPD; n=57, 57 | 66.2 (8.66) | 66.7 (8.70)
  Asthma; n=33, 33 | 64.8 (8.99) | 65.7 (9.49)
  COPD; n=24, 24 | 68.2 (7.96) | 68.1 (7.45)

14. Secondary Outcome: Mean of Maximum Heart Rate Over 0 to 4 Hours Post Dose for Salmeterol
Description: The maximum observed value of heart rate was measured from the time of the morning dose on Day 10 to 4 hours post dose.
Time Frame: as for outcome 13
Population: PK/PD Population
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
bpm
  Asthma + COPD; n=57, 57 | 73.0 (9.86) | 74.3 (9.08)
  Asthma; n=33, 33 | 72.3 (10.52) | 73.5 (9.62)
  COPD; n=24, 24 | 74.0 (8.98) | 75.4 (8.35)

15. Secondary Outcome: Minimum Diastolic Blood Pressure (DBP), Maximum Systolic Blood Pressure (SBP), and Weighted Mean for DBP and SBP Over 0 to 4 Hours Post Dose
Description: The diastolic and systolic blood pressure of the participants was measured. The maximum and minimum observed values from the time of the morning dose on Day 10 to 4 hours post dose were measured for SBP and DBP. The weighted mean value from the time of the morning dose on Day 10 to 4 hours post dose was calculated. Weighted mean was calculated by using all values of DBP and SBP at the indicated timepoint contributing to the calculation of the mean but with different weightage.
Time Frame: as for outcome 13
Population: PK/PD Population
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
millimeters of mercury (mmHg)
  DBP, Asthma + COPD; n=57, 57 | 64.7 (8.16) | 66.2 (8.12)
  DBP, Asthma; n=33, 33 | 61.6 (6.66) | 62.6 (5.27)
  DBP, COPD; n=24, 24 | 69.1 (8.14) | 71.2 (8.83)
  Weighted mean DBP, Asthma + COPD; n=57, 57 | 71.1 (7.85) | 72.2 (8.13)
  Weighted mean DBP, Asthma; n=33, 33 | 68.0 (5.69) | 68.8 (5.26)
  Weighted mean DBP, COPD; n=24, 24 | 75.4 (8.18) | 77.0 (9.04)
  SBP, Asthma + COPD; n=57, 57 | 128.0 (14.26) | 129.3 (13.63)
  SBP, Asthma; n=33, 33 | 119.9 (8.25) | 122.1 (9.08)
  SBP, COPD; n=24, 24 | 139.1 (13.29) | 139.1 (12.82)
  Weighted mean SBP, Asthma + COPD; n=57, 57 | 118.8 (11.78) | 120.3 (11.69)
  Weighted mean SBP, Asthma; n=33, 33 | 112.9 (7.97) | 114.6 (8.25)
  Weighted mean SBP, COPD; n=24, 24 | 126.9 (11.44) | 128.2 (11.21)

16. Secondary Outcome: Maximum and Weighted Mean Over 0 to 4 Hours Post Dose of the QT Interval Corrected According to Bazett's Formula (QTc[B]) and the QT Interval Corrected According to Fridericia's Formula (QTc[F])
Description: The electrocardiogram (ECG) of the participants was taken, and the maximum and weighted mean of QTc(B) and QTc(F) was measured. Weighted mean was calculated by using all values of QTc(B) and QTc(F) at the indicated timepoint contributing to the calculation of the mean but with different weightage. The ECG helps in the assessment of the condition of the heart. The QT interval gives the measure of the heart rate, and the cQT interval gives the corrected value.
Time Frame: At pre-morning dose; 15, 30, 60, 90 minutes post-dose (PD); and 2, 3 and 4 hours PD on Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: PK/PD Population
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
Milliseconds (msec)
  Max, QTc(B) interval, Asthma + COPD; n=57, 57 | 434.0 (22.49) | 434.4 (25.39)
  Max, QTc(B) interval, Asthma; n=33, 33 | 423.7 (18.22) | 424.7 (19.86)
  Max, QTc(B) interval, COPD; n=24, 24 | 448.1 (20.29) | 447.6 (26.53)
  Weighted mean QTc(B), Asthma + COPD; n=57, 57 | 416.8 (23.24) | 416.8 (24.23)
  Weighted mean QTc(B), Asthma; n=33, 33 | 405.7 (18.61) | 406.3 (20.81)
  Weighted mean QTc(B), COPD; n=24, 24 | 431.9 (20.48) | 431.3 (21.25)
  Max QTc(F), Asthma + COPD; n=57, 57 | 422.5 (19.31) | 422.6 (22.43)
  Max QTc(F), Asthma; n=33, 33 | 413.5 (15.01) | 413.7 (17.52)
  Max QTc(F), COPD; n=24, 24 | 434.9 (17.83) | 434.9 (22.96)
  Weighted mean QTc(F), Asthma + COPD; n=57, 57 | 410.3 (19.34) | 410.1 (20.28)
  Weighted mean QTc(F), Asthma; n=33, 33 | 401.2 (15.03) | 401.3 (17.13)
  Weighted mean QTc(F), COPD; n=24, 24 | 422.9 (17.63) | 422.3 (18.06)

17. Secondary Outcome: Weighted Mean Over 0 to 4 Hours Post Dose of Plasma Potassium and Minimum (Min) Plasma Potassium
Description: Blood samples of participants were collected for the evaluation of weighted mean over 0 to 4 hours post dose and the minimum plasma potassium level. Weighted mean was calculated by using all values of plasma potassium at the indicated timepoint contributing to the calculation of the mean but with different weightage.
Time Frame: At pre-morning dose; 30, 60 minutes post-dose (PD); and 2 and 4 hours PD on Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
Millimoles per liter (mmol/L)
  Weighted mean, Asthma + COPD; n=56, 57 | 4.11 (0.209) | 4.11 (0.228)
  Weighted mean, Asthma; n=32, 33 | 4.11 (0.216) | 4.10 (0.242)
  Weighted mean, COPD; n=24, 24 | 4.11 (0.204) | 4.13 (0.210)
  Min, Asthma + COPD; n=57, 57 | 3.91 (0.231) | 3.90 (0.249)
  Min, Asthma; n=33, 33 | 3.92 (0.241) | 3.89 (0.269)
  Min, COPD; n=24, 24 | 3.89 (0.220) | 3.92 (0.221)

18. Secondary Outcome: Weighted Mean Over 0 to 4 Hours Post Dose and Maximum Plasma Glucose
Description: Blood samples of participants were collected for the evaluation of weighted mean over 0 to 4 hours post dose and the maximum plasma glucose level. Weighted mean was calculated by using all values of plasma glucose at the indicated timepoint contributing to the calculation of the mean but with different weightage.
Time Frame: as for outcome 17
Population: PK/PD Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 57 | 57
mmol/L
  Weighted mean, Asthma + COPD; n=57, 57 | 5.85 (1.119) | 5.95 (0.999)
  Weighted mean, Asthma; n=33, 33 | 5.67 (0.622) | 5.80 (0.654)
  Weighted mean, COPD; n=24, 24 | 6.11 (1.545) | 6.16 (1.325)
  Max, Asthma + COPD; n=57, 57 | 6.94 (1.644) | 7.19 (1.614)
  Max, Asthma; n=33, 33 | 6.64 (1.147) | 6.96 (1.125)
  Max, COPD; n=24, 24 | 7.36 (2.105) | 7.50 (2.098)

19. Secondary Outcome: Mean Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, and White Blood Cell (WBC) Count
Description: Blood samples of participants were collected for the evaluation of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count, and WBC count. Data are reported for the first (1st) and second (2nd) administration (admin) of FP/salmeterol via MDPI or capsule-based inhaler. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: Day 10 of each study period (P): Study Day (SD) 10 (reference day is SD 1 or Randomization day), 20, 30, and 40 (+/-1) for P 1, 2, 3, and 4, respectively
Population: All Subjects Population: all participants who received at least one dose of study medication. Out of the total population, 34 participants had asthma and 26 participants had COPD. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells/L
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
Giga (10^9) cells/L
  Basophils, 1st admin, Asthma; n=33, 33 | 0.05 (0.051) | 0.06 (0.082)
  Basophils, 2nd admin, Asthma; n=31, 33 | 0.04 (0.050) | 0.04 (0.050)
  Basophils, 1st admin, COPD; n=25, 25 | 0.07 (0.085) | 0.04 (0.050)
  Basophils, 2nd admin, COPD; n=24, 25 | 0.04 (0.050) | 0.04 (0.050)
  Eosinophils, 1st admin, Asthma; n=33, 33 | 0.37 (0.238) | 0.33 (0.187)
  Eosinophils, 2nd admin, Asthma; n=31, 33 | 0.31 (0.182) | 0.31 (0.189)
  Eosinophils, 1st admin, COPD; n=25, 25 | 0.25 (0.169) | 0.23 (0.173)
  Eosinophils, 2nd admin, COPD; n=24, 25 | 0.25 (0.169) | 0.26 (0.171)
  Lymphocytes, 1st admin, Asthma; n=33, 33 | 1.96 (0.497) | 1.92 (0.454)
  Lymphocytes, 2nd admin, Asthma; n=31,33 | 1.90 (0.461) | 1.86 (0.478)
  Lymphocytes, 1st admin, COPD; n=25, 25 | 1.70 (0.419) | 1.72 (0.472)
  Lymphocytes, 2nd admin, COPD; n=24, 25 | 1.75 (0.475) | 1.68 (0.352)
  Monocytes, 1st admin, Asthma; n=33, 33 | 0.54 (0.162) | 0.55 (0.175)
  Monocytes, 2nd admin, Asthma; n=31, 33 | 0.54 (0.133) | 0.52 (0.156)
  Monocytes, 1st admin, COPD; n=25, 25 | 0.64 (0.161) | 0.60 (0.181)
  Monocytes, 2nd admin, COPD; n=24, 25 | 0.63 (0.157) | 0.63 (0.170)
  TN, 1st admin, Asthma; n=33, 33 | 3.28 (1.097) | 3.37 (1.036)
  TN, 2nd admin, Asthma; n=31, 33 | 3.30 (0.904) | 3.28 (1.083)
  TN, 1st admin, COPD; n=25, 25 | 3.70 (1.601) | 3.48 (1.059)
  TN, 2nd admin, COPD; n=24, 25 | 3.45 (1.060) | 3.75 (1.595)
  Platelet count, 1st admin, Asthma; n=33, 33 | 225.1 (40.05) | 223.9 (41.64)
  Platelet count, 2nd admin, Asthma; n=31, 33 | 230.7 (43.08) | 230.8 (49.90)
  Platelet count, 1st admin, COPD; n=24, 24 | 230.6 (50.56) | 226.6 (52.85)
  Platelet count, 2nd admin, COPD; n=23, 24 | 235.1 (52.73) | 240.1 (48.78)
  WBC count, 1st admin, Asthma; n=33, 33 | 6.145 (1.3253) | 6.182 (1.3646)
  WBC count, 2nd admin, Asthma; n=31, 33 | 6.071 (1.1892) | 5.976 (1.3528)
  WBC count, 1st admin, COPD; n=25, 25 | 6.340 (1.9346) | 6.036 (1.3076)
  WBC count, 2nd admin, COPD; n=24, 25 | 6.092 (1.2752) | 6.312 (1.8600)

20. Secondary Outcome: Mean Hemoglobin and Mean Corpuscular Hemoglobin (MCH) Concentration
Description: Blood samples of participants were collected for the evaluation of mean hemoglobin (mean level of hemoglobin in the whole blood sample) and MCH concentration. The MCH concentration is the average concentration of hemoglobin in a red blood cell. Hemoglobin is the red pigment in the blood, and it is reponsible for carrying oxygen. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: All Subjects Population. Out of the total population, 34 participants had asthma and 26 participants had COPD. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
Grams per liter (g/L)
  Hemoglobin, 1st admin, Asthma; n=33, 33 | 138.2 (12.20) | 135.4 (12.32)
  Hemoglobin, 2nd admin, Asthma; n=31, 33 | 133.0 (14.31) | 132.3 (13.44)
  Hemoglobin, 1st admin, COPD; n=25, 25 | 133.3 (12.07) | 133.1 (11.66)
  Hemoglobin, 2nd admin, COPD; n=24, 25 | 130.6 (14.65) | 128.5 (14.14)
  MCH concentration, 1st admin, Asthma; n=33, 33 | 334.7 (9.85) | 334.0 (10.38)
  MCH concentration, 2nd admin, Asthma; n=31, 33 | 333.0 (11.21) | 333.2 (10.92)
  MCH concentration, 1st admin, COPD; n=,25, 25 | 329.0 (9.69) | 328.5 (9.37)
  MCH concentration, 1st admin, COPD; n=24, 25 | 327.4 (11.47) | 328.8 (11.33)

21. Secondary Outcome: Red Blood Cell (RBC) Count and Reticulocytes
Description: Blood samples of participants were collected for the evaluation of RBC and reticulocytes count. Reticulocytes are immature red blood cells. Normally, about 1% to 2% of the red blood cells in the blood are reticulocytes. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Trillion (10^12) cells/L
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
Trillion (10^12) cells/L
  RBC, 1st admin, Asthma; n=33, 33 | 4.608 (0.3590) | 4.542 (0.3616)
  RBC, 2nd admin, Asthma; n=31, 33 | 4.460 (0.4059) | 4.424 (0.3638)
  RBC, 1st admin, Asthma, COPD; n=25, 25 | 4.523 (0.5483) | 4.530 (0.5906)
  RBC, 2nd admin, COPD; n=24, 25 | 4.438 (0.6062) | 4.358 (0.6342)
  Reticulocytes, 1st admin, Asthma ; n=33, 32 | 0.049 (0.0178) | 0.050 (0.0168)
  Reticulocytes, 2nd admin, Asthma; n=31, 33 | 0.051 (0.0195) | 0.050 (0.0193)
  Reticulocytes, 1st admin, COPD; n=25, 25 | 0.054 (0.0191) | 0.054 (0.0230)
  Reticulocytes, 2nd admin, COPD; n=24, 25 | 0.059 (0.0252) | 0.061 (0.0271)

22. Secondary Outcome: Mean Corpuscule Hemoglobin (MCH)
Description: Blood samples of participants were collected for the evaluation of MCH. MCH is the average mass or amount of hemoglobin per red blood cell in a sample of blood. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: All Subject Population. Out of the total population, 34 participants had asthma and 26 participants had COPD. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: picograms (pg)/cell
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
picograms (pg)/cell
  1st admin, Asthma; n=33, 33 | 29.99 (1.422) | 29.86 (1.399)
  2nd admin, Asthma; n=31, 33 | 29.80 (1.501) | 29.92 (1.456)
  1st admin, COPD; n=25, 25 | 29.72 (2.920) | 29.72 (2.945)
  2nd admin, COPD; n=24, 25 | 29.73 (3.079) | 29.83 (2.993)

23. Secondary Outcome: Mean Corpuscle Volume (MCV)
Description: Blood samples of participants were collected for the evaluation of MCV. MCV is a measure of the average red blood cell size that is reported as part of a standard complete blood count. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Femtoliters (fL; 10^-15 L)/cell
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
Femtoliters (fL; 10^-15 L)/cell
  1st admin, Asthma; n=33, 33 | 89.65 (2.808) | 89.41 (2.862)
  2nd admin, Asthma; n=31, 33 | 89.52 (2.953) | 89.77 (2.821)
  1st admin, COPD; n=25, 25 | 90.21 (7.643) | 90.37 (7.595)
  2nd admin, COPD; n=24, 25 | 90.76 (7.609) | 90.64 (7.498)

24. Secondary Outcome: Mean Hematocrit
Description: Blood samples of participants were collected for the evaluation of hematocrit. The hematocrit is the percentage of the RBCs in the blood. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of RBCs
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
percentage of RBCs
  1st admin, Asthma; n=33, 33 | 0.413 (0.0318) | 0.405 (0.0328)
  2nd admin, Asthma; n=31, 33 | 0.399 (0.0375) | 0.396 (0.0345)
  1st admin, COPD; n=25, 25 | 0.405 (0.0346) | 0.405 (0.0379)
  2nd admin, COPD; n=24, 25 | 0.400 (0.0448) | 0.391 (0.0441)

25. Secondary Outcome: Mean Albumin and Total Protein
Description: The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
g/L
  Albumin, 1st admin, Asthma; n=33, 33 | 43.0 (2.47) | 42.3 (2.16)
  Albumin, 2nd admin, Asthma; n=31, 33 | 42.0 (2.02) | 41.8 (2.77)
  Albumin, 1st admin, COPD; n=25, 25 | 40.9 (2.19) | 41.4 (2.08)
  Albumin, 2nd admin, COPD; n=25, 25 | 40.8 (2.30) | 40.0 (2.12)
  Total protein, 1st admin, Asthma; n=33, 33 | 66.8 (4.29) | 66.0 (3.24)
  Total protein, 2nd admin, Asthma; n=31, 33 | 65.4 (3.48) | 64.8 (4.68)
  Total protein, 1st admin, COPD; n=25, 25 | 64.7 (3.82) | 64.9 (4.16)
  Total protein, 2nd admin, COPD; n=25, 25 | 64.6 (4.01) | 63.5 (4.00)

26. Secondary Outcome: Mean Alkaline Phosphatase (AP), Alanine Amino Transferase (ALT), Aspartate Amio Transferase (AST), and Gama Glutamyl Transferase (GGT)
Description: Blood samples of participants were collected for the evaluation of AP, ALT, AST, and GGT. All of these parameters are measured to help assess the condition of the liver. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
International units per liter (IU/L)
  AP, 1st admin, Asthma; n=33, 33 | 64.6 (15.00) | 63.4 (14.30)
  AP, 2nd admin, Asthma; n=31, 33 | 65.0 (14.87) | 63.9 (15.74)
  AP, 1st admin, COP ; n=25, 25 | 69.6 (20.28) | 69.9 (22.14)
  AP, 2nd admin, COPD; n=25, 25 | 69.8 (18.31) | 68.4 (17.78)
  ALT, 1st admin, Asthma; n=33, 33 | 20.1 (9.49) | 20.4 (8.68)
  ALT, 2nd admin, Asthma; n=31, 33 | 21.5 (11.32) | 19.1 (8.21)
  ALT, 1st admin, COPD; n=25, 25 | 21.2 (10.47) | 23.4 (15.45)
  ALT, 2nd admin, COPD; n=25, 25 | 20.9 (10.80) | 21.2 (10.33)
  AST, 1st admin, Asthma; n=33, 33 | 21.2 (8.22) | 21.6 (4.42)
  AST, 2nd admin, Asthma; n=31, 33 | 20.7 (5.85) | 20.1 (4.87)
  AST, 1st admin, COPD; n=25, 25 | 22.7 (7.44) | 24.7 (14.22)
  AST, 2nd admin, COPD; n=25, 25 | 22.5 (8.95) | 21.1 (7.82)
  GGT, 1st admin, Asthma; n=33, 33 | 21.3 (14.51) | 21.0 (15.18)
  GGT, 2nd admin, Asthma; n=31, 33 | 22.7 (19.22) | 21.0 (15.06)
  GGT, 1st admin, COPD; n=25, 25 | 36.9 (53.90) | 44.0 (80.65)
  GGT, 2nd admin, COPD; n=25, 25 | 31.8 (32.85) | 29.6 (24.43)

27. Secondary Outcome: Mean Direct Bilirubin (DB), Total Bilirubin (TB), Creatinine, and Uric Acid
Description: Blood samples of participants were collected for the evaluation of DP, TB, creatinine, and uric acid. DB and TB are measures that help assess the condition of the liver, and creatinine and uric acid are measures that help assess the condition of the kidneys. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
Micromoles per liter (µmol/L)
  DB, 1st admin, Asthma; n=33, 33 | 3.2 (2.83) | 2.7 (1.99)
  DB, 2nd admin, Asthma; n=31, 33 | 3.0 (1.47) | 2.6 (1.11)
  DB, 1st admin, COPD; n=25, 25 | 2.9 (0.97) | 2.8 (1.05)
  DB, 2nd admin, COPD; n=25, 25 | 2.7 (1.16) | 2.9 (1.22)
  TB, 1st admin, Asthma; n=33, 33 | 9.5 (3.58) | 9.9 (5.12)
  TB, 2nd admin, Asthma; n=31, 33 | 9.9 (4.48) | 8.6 (3.57)
  TB, 1st admin, COPD; n=25, 25 | 8.7 (2.42) | 9.4 (3.67)
  TB, 2nd admin, COPD; n=25, 25 | 8.5 (2.76) | 8.4 (3.51)
  Creatinine, 1st admin, Asthma; n=33, 33 | 77.2 (11.48) | 75.8 (11.04)
  Creatinine, 2nd admin, Asthma; n=31, 33 | 76.9 (10.81) | 75.2 (11.39)
  Creatinine, 1st admin, COPD; n=25, 25 | 79.4 (18.33) | 77.7 (16.45)
  Creatinine, 2nd admin, COPD; n=25, 25 | 79.6 (17.38) | 79.4 (18.45)
  Uric acid, 1st admin, Asthma n=33, 33 | 328.9 (73.11) | 331.5 (66.84)
  Uric acid, 2nd admin, Asthma; n=31, 33 | 338.4 (67.25) | 325.6 (70.04)
  Uric acid, 1st admin, COPD; n=25, 25 | 354.2 (60.13) | 348.3 (59.25)
  Uric acid, 2nd admin, COPD; n=25, 25 | 361.7 (65.96) | 352.0 (64.39)

28. Secondary Outcome: Mean Calcium, Chloride, Glucose, Potassium, Sodium, Carbon Dioxide (CO2) Content/Bicarbonate (Bicar), and Urea/Blood Urea Nitrogen (BUN)
Description: Blood samples of participants were collected for the evaluation of calcium, chloride, glucose, potassium, sodium, carbon dioxide (CO2) content/bicarbonate, and urea/BUN. All of these parameters are measured to help assess the condition of the kidneys. The timing of the first and second administrations depended on the randomization schedule. If the treatment sequence received was "ABBA," then Days 10 and 40, respectively, correspond to the first and second administrations for treatment A.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 33
µmol/L
  Calcium, 1st admin, Asthma; n=33, 32 | 2.191 (0.0954) | 2.178 (0.0900)
  Calcium, 2nd admin, Asthma; n=31, 33 | 2.190 (0.0799) | 2.170 (0.1382)
  Calcium, 1st admin, COPD; n=25, 25 | 2.205 (0.0874) | 2.189 (0.0946)
  Calcium, 2nd admin, COPD; n=25, 25 | 2.206 (0.0998) | 2.190 (0.0916)
  Chloride, 1st admin, Asthma; n=33, 33 | 104.7 (2.38) | 104.8 (2.28)
  Chloride, 2nd admin, Asthma; n=31, 33 | 104.5 (2.29) | 105.3 (2.89)
  Chloride, 1st admin, COP; n=25, 25 | 104.4 (2.80) | 104.0 (2.67)
  Chloride, 2nd admin, COPD n=25, 25 | 104.1 (2.49) | 104.4 (2.90)
  Glucose, 1st admin, Asthma; n=33, 33 | 5.06 (0.555) | 5.06 (0.445)
  Glucose, 2nd admin, Asthma; n=31, 33 | 5.06 (0.325) | 5.15 (0.484)
  Glucose, 1st admin, COPD; n=25, 25 | 5.36 (0.846) | 5.37 (1.306)
  Glucose, 2nd admin, COPD; n=25, 25 | 5.63 (1.143) | 5.45 (0.856)
  Potassium, 1st admin, Asthma; n=32, 33 | 4.15 (0.421) | 4.05 (0.271)
  Potassium, 2nd admin, Asthma; n=31, 33 | 4.06 (0.291) | 4.02 (0.269)
  Potassium, 1st admin, COPD n=25, 25 | 4.16 (0.212) | 4.08 (0.233)
  Potassium, 2nd admin, COPD; n=25, 25 | 4.10 (0.223) | 4.11 (0.272)
  Sodium, 1st admin, Asthma; n=33, 33 | 140.5 (1.80) | 140.5 (1.60)
  Sodium, 2nd admin, Asthma; n=31, 33 | 140.1 (2.13) | 140.4 (1.34)
  Sodium, 1st admin, COPD n=25, 25 | 140.5 (2.69) | 140.5 (2.96)
  Sodium, 2nd admin, COPD n=25, 25 | 140.1 (2.49) | 140.2 (2.59)
  CO2 content/bicar, 1st admin, Asthma; n=33, 33 | 26.1 (2.09) | 25.6 (2.26)
  CO2 content/bicar, 2nd admin, Asthma; n=31, 33 | 26.2 (2.22) | 26.0 (2.58)
  CO2 content/bicar, 1st admin, COPD; n=25, 25 | 27.2 (1.90) | 27.3 (1.89)
  CO2 content/bicar, 2nd admin, COPD; n=25, 25 | 27.3 (2.08) | 27.2 (1.89)
  Urea/BUN, 1st admin, Asthma; n=33, 33 | 5.34 (1.389) | 5.41 (1.406)
  Urea/BUN, 2nd admin, Asthma; n=31, 33 | 5.31 (1.290) | 5.43 (1.312)
  Urea/BUN, 1st admin, COPD; n=25, 25 | 5.98 (1.426) | 6.09 (1.473)
  Urea/BUN, 2nd admin, COPD; n=25, 25 | 5.90 (1.402) | 6.12 (1.446)

29. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Randomization (Day 1) up to Follow-up (Days 47-50)
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | FP/Salmeterol From MDPI | FP/Salmeterol From Capsule-based Inhaler
Number analyzed (Participants) | 33 | 34
participants
  1st admin, Asthma; n=33, 34 | 13 | 13
  2nd admin, Asthma; n=31, 33 | 12 | 15
  1st admin, COPD; n=26, 25 | 14 | 11
  2nd admin, COPD; n=25, 25 | 9 | 11

ADVERSE EVENTS:
Groups:
- FP/Salmeterol From MDPI 1st Administration (Admin), Asthma: Fluticasone propionate (FP)/salmeterol combination was administered to participants with asthma as a powder in blister in the dose of 250/50 micrograms (mcg) twice daily (BID) via a multi-dose dry powder inhaler (MDPI) for a 10-day period.
- FP/Salmeterol From MDPI 2nd Admin, Asthma: Fluticasone propionate (FP)/salmeterol combination was administered to particiapants with asthma as a powder in blister in the dose of 250/50 micrograms (mcg) twice daily (BID) via a multi-dose dry powder inhaler (MDPI) for a 10-day period.
- FP/Salmeterol From Capsule-based Inhaler 1st Admin, Asthma; FP/Salmeterol From Capsule-based Inhaler 2nd Admin, Asthma: Fluticasone propionate (FP)/salmeterol combination was administered to participants with asthma as a powder in capsule in the dose of 250/50 mcg BID via a capsule-based inhaler for a 10-day period.
- FP/Salmeterol From MDPI 1st Admin, COPD; FP/Salmeterol From MDPI 2nd Admin, COPD: Fluticasone propionate (FP)/salmeterol combination was administered to participants with COPD as a powder in blister in the dose of 250/50 micrograms (mcg) twice daily (BID) via a multi-dose dry powder inhaler (MDPI) for a 10-day period.
- FP/Salmeterol From Capsule-based Inhaler 1st Admin, COPD; FP/Salmeterol From Capsule-based Inhaler 2nd Admin, COPD: Fluticasone propionate (FP)/salmeterol combination was administered to participants with COPD as a powder in capsule in the dose of 250/50 mcg BID via a capsule-based inhaler for a 10-day period.
Arm/Group | FP/Salmeterol From MDPI 1st Administration (Admin), Asthma | FP/Salmeterol From MDPI 2nd Admin, Asthma | FP/Salmeterol From Capsule-based Inhaler 1st Admin, Asthma | FP/Salmeterol From Capsule-based Inhaler 2nd Admin, Asthma | FP/Salmeterol From MDPI 1st Admin, COPD | FP/Salmeterol From MDPI 2nd Admin, COPD | FP/Salmeterol From Capsule-based Inhaler 1st Admin, COPD | FP/Salmeterol From Capsule-based Inhaler 2nd Admin, COPD
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31 | 0/34 | 1/33 | 0/26 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 13/33 | 12/31 | 13/34 | 15/33 | 14/26 | 9/25 | 11/25 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP/Salmeterol From MDPI 1st Administration (Admin), Asthma (N=33) | FP/Salmeterol From MDPI 2nd Admin, Asthma (N=31) | FP/Salmeterol From Capsule-based Inhaler 1st Admin, Asthma (N=34) | FP/Salmeterol From Capsule-based Inhaler 2nd Admin, Asthma (N=33) | FP/Salmeterol From MDPI 1st Admin, COPD (N=26) | FP/Salmeterol From MDPI 2nd Admin, COPD (N=25) | FP/Salmeterol From Capsule-based Inhaler 1st Admin, COPD (N=25) | FP/Salmeterol From Capsule-based Inhaler 2nd Admin, COPD (N=25)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP/Salmeterol From MDPI 1st Administration (Admin), Asthma (N=33) | FP/Salmeterol From MDPI 2nd Admin, Asthma (N=31) | FP/Salmeterol From Capsule-based Inhaler 1st Admin, Asthma (N=34) | FP/Salmeterol From Capsule-based Inhaler 2nd Admin, Asthma (N=33) | FP/Salmeterol From MDPI 1st Admin, COPD (N=26) | FP/Salmeterol From MDPI 2nd Admin, COPD (N=25) | FP/Salmeterol From Capsule-based Inhaler 1st Admin, COPD (N=25) | FP/Salmeterol From Capsule-based Inhaler 2nd Admin, COPD (N=25)
Headache (Nervous system disorders) | 8 | 7 | 10 | 10 | 5 | 5 | 2 | 3
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.